CLINICAL TRIAL: NCT01038843
Title: A Randomised, Double-blind, Placebo-controlled, Parallel Group, Dose-titration Study to Determine the Efficacy and Safety of VA106483 in Male Subjects With Nocturia
Brief Title: Efficacy Study of VA106483 in Males With Nocturia.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Vantia Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 483-005
Record Dates: First submitted 2009-12-22; First posted 2009-12-24 (Estimated); Last update posted 2014-06-20 (Estimated); Status verified 2014-06

CONDITIONS: Nocturia
Keywords: VA106483; Nocturia; males; nocturnal voids; anti-diuretic; hyponatraemia
MeSH Terms: conditions — Nocturia; Hyponatremia

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- VA106483 1mg (Experimental)
  Interventions: Drug: VA106483
- VA106483 2mg (Experimental)
  Interventions: Drug: VA106483
- VA106483 4mg (Experimental)
  Interventions: Drug: VA106483
- Sugar pill (Placebo Comparator)
  Interventions: Drug: VA106483

INTERVENTIONS:
Drug: VA106483 — Drug: VA106483 Once daily oral dose of 1 mg VA106483 or matching placebo for 14 (+3) days. Once daily oral dose of 2 mg VA106483 or matching placebo for 14 (+3) days. Once daily oral dose of 4 mg VA106483 or matching placebo for 28 days.
  Placebo: as above

SUMMARY:
To investigate the effect of VA106483 on nocturia related clinical outcomes compared to placebo.

DETAILED DESCRIPTION:
Nocturia, defined as waking to urinate at least once per night between periods of sleep, is a common complaint which increases with age. VA106483 is a non-peptide drug VA106483 that is being developed for the treatment of nocturia in males.

The purpose of this study is to investigate the effect of VA106483 on the number of times the subject needs to get up to urinate (nocturnal void) per night and to determine the effect on the time between the subject's bedtime and the time they first wake up to urinate.

ELIGIBILITY:
Inclusion Criteria:

* Male subjects aged ≥18 years (no upper limit) with nocturia
* Generally well (concomitant illness/conditions well controlled)
* Serum sodium within the normal limits
* Normal or not clinically significant prostate specific antigen levels
* Able to comply with the requirements of the study
* Provide written informed consent

Exclusion Criteria:

* Prostatic cancer
* Signs or symptoms of heart failure
* Peripheral pitting oedema extending ≥10 cm above the ankle
* Palpable bladder or pelvic mass on abdominal examination
* Enuresis or night-time incontinence
* Excessive nocturnal void frequency
* Sleep disorders
* Diabetes insipidus or uncontrolled diabetes mellitus
* Presence of blood or glucose in the urine on urinalysis that is clinically significant
* Urinary tract infection
* Polydipsia
* Syndrome of inappropriate antidiuretic hormone secretion
* Body mass index ≥35
* High calcium levels or low potassium levels
* Other protocol defined eligibility criteria may apply

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 152 (Actual)
Dates: Start 2009-12; Primary Completion 2010-07 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
Change in the mean number of nocturnal voids per night | 70 days

SECONDARY OUTCOMES:
Mean duration of first sleep period | 70 days
Change in nocturia-related quality of life | 70 days
Incidence and frequency of adverse events | 70 days
Frequency of hyponatraemia | 70 days
Change from baseline in safety laboratory parameters | 70 days

CONTACTS AND LOCATIONS:
Overall Officials: Mira Baron, Principal Investigator — Rapid Medical Research, Inc.; David Beccia, Principal Investigator — Medical & Clinical Research Associates; Kenneth Blaze, Principal Investigator — South Broward Research, LLC; Mitchell Efros, Principal Investigator — Accumed Research Associates; Marc Gittelman, Principal Investigator — South Florida Medical Research; Evan Goldfischer, Principal Investigator — Hudson Valley Urology, PC; Elizabeth Houser, Principal Investigator — The Urology Team P.A.; Theodore Johnson II, Principal Investigator — Emory University; Steven Kester, Principal Investigator — Urology Center of Florida; Richard Lotenfoe, Principal Investigator — Discovery Clinical Trials; Earl Martin, Principal Investigator — Martin Diagnostic Clinic; H. David Mitcheson, Principal Investigator — Bay State Clinical Trials, Inc.; Chris Ng, Principal Investigator — Tower Urology Medical Group; Aris Nikas, Principal Investigator — Health Texas Research Institute; Joseph Parkhurst, Principal Investigator — Parkhurst Research Organization; Bruce Rankin, Principal Investigator — Avail Clinical Research LLC; Leah Schmidt, Principal Investigator — Genova Clinical Research; Howard Hezmall, Principal Investigator — Urology Associates of North Texas; Wilbur Wells Jnr, Principal Investigator — Alabama Research Center, LLC; Rafael Wurzel, Principal Investigator — Grove Hill Clinical Research
Locations (19):
- United States (19):
  - Alabama Research Center, LLC, Birmingham, Alabama
  - Genova Clinical Research, Tucson, Arizona
  - Tower Urology Medical Group, Los Angeles, California
  - Grove Hill Clinical Research, New Britian, Connecticut
  - South Florida Medical Research, Aventura, Florida
  - Discovery Clinical Trials, Celebration, Florida
  - Avail Clinical Research LLC, DeLand, Florida
  - Urology Center of Florida, Hialeah, Florida
  - South Broward Research, LLC, Pembroke Pines, Florida
  - Bay State Clinical Trials, Inc., Watertown, Massachusetts
  - Medical & Clinical Research Associates, Bay Shore, New York
  - Accumed Research Associates, Garden City, New York
  - Hudson Valley Urology, PC, Poughkeepsie, New York
  - Rapid Medical Research, Inc., Clevland, Ohio
  - Parkhurst Research Organization, Bethany, Oklahoma
  - Urology Associates of North Texas, Arlington, Texas
  - The Urology Team P.A., Austin, Texas
  - Health Texas Research Institute, San Antonio, Texas
  - Martin Diagnostic Clinic, Tomball, Texas